CLINICAL TRIAL: NCT05835934
Title: A Phase I Clinical Study on Absorption, Metabolism, and Excretion of [14C]HSK21542 in Healthy Adult Male Chinese Subjects - Mass Balance and Biotransformation of [14C]HSK21542 in Human.
Brief Title: Pharmacokinetics, Mass Balance, and Metabolism of [14C]HSK21542 in Healthy Adult Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK21542-103
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Analgesic and Anti-itch

STUDY DESIGN:
Intervention Model Description: A single-center, single-dose, non-randomized, open-label design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental): 2 μg/0.212 μCi/kg [14C]HSK21542
  Interventions: Drug: [14C]HSK21542

INTERVENTIONS:
Drug: [14C]HSK21542 — A single intravenous dose of 2 μg/0.212 μCi/kg [14C]HSK21542 in boluses within 2 minute after fasting for at least 10 hours.

SUMMARY:
This is a single-center, nonrandomized, and open design study to investigate the pharmacokinetics, mass balance, metabolism and excretion of HSK21542 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese males, aged 18-45 years old (inclusive);
2. Body weight ≥ 50.0 kg and body mass index (BMI) between 19.0-26.0 kg/m2 (inclusive);
3. Vital signs: blood pressure between 90-139/60-89 mmHg; heart rate or pulse between 60-99 beats/min;
4. Subjects judged by the investigator based on past medical history, comprehensive physical examination, vital signs examination, and other prescribed tests;
5. Subjects who voluntarily sign the informed consent form (ICF), able to communicate with the investigator and to complete all trial procedures as per the protocol.

Exclusion Criteria:

1. Clinically significant abnormal results for comprehensive physical examination, vital signs, routine laboratory tests [blood routine, blood biochemistry, coagulation routine, urine routine, stool routine + occult blood, thyroid function, visual acuity and ophthalmic examination (slit lamp, introcular pressure, and fundoscopy), 12-lead electrocardiogram (ECG), chest X-ray (anteriorposterior), and abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, and kidney);
2. Positive for hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody, or Treponema pallidum antibodies;

   Medication history:
3. Use of any Western medicine or Chinese patent medicine (including prescription drug, over-the-counter drug, health care product, or live attenuated influenza vaccine) within 14 days prior to screening;
4. Participation in any clinical trial and interference with other investigational drug or medical device within 3 month prior to screening;

   Medical history and surgical history:
5. History of serious clinical diseases or diseases/conditions that the investigator believes may affect the study results, including but not limited to the history of diseases in the motor system, nervous system, endocrine system, circulatory system, respiratory system, digestive system, urinary system, and reproductive system;
6. Past history of organic heart disease, heart failure, myocardial infarction, angina, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, long QT syndrome or symptoms and familial history of long QT syndrome (indicated by genetic evidence or sudden death of a close relative at a young age due to cardiac causes);
7. Have undergone major surgery within 6 months prior to screening or with incomplete healing of the surgical incision; major surgery includes, but is not limited to, any surgery with significant risk of bleeding, prolonged general anesthesia, or incisional biopsy or obvious traumatic injury (excluding cured appendicitis surgery or rectal prolapse surgery);
8. Severe allergic constitution, including known allergy to any excipient of this investigational product (Glacial acetic acid, sodium acetate, water for injection), two or more drugs and food components, or with special dietary requirements and thus unable to follow a standardized diet;

   Living habits:
9. Long-term excessive consumption (more than 8 cups a day, 1 cup =250mL) of tea, grapefruit, coffee, drinks containing caffeine or grapefruit;
10. Subjects with a history of alcohol abuse in the three months prior to screening, with an average daily intake of more than 15 g of alcohol (15 g of alcohol is equivalent to 360 mL of beer or 150 mL of wine or 50 mL of liquor containing 40% alcohol), or with a positive alcohol breath test (test value greater than 20 mg/100 mL);
11. Subjects who smoked more than 5 cigarettes a day or habitually used nicotine-containing products in the 3 months before the screening period and could not quit during the test period;
12. Drug abuse or dependence, urine screening positive for drug abuse;

    Others:
13. Workers engaged in work requiring prolonged exposure to radioactivity; Or had significant radiation exposure (≥2 chest/abdominal CT scans, or ≥3 other types of X-rays) within 1 year or participated in the radiopharma labeling test prior to the test;
14. Those who had a birth plan during the study period and within 1 year after completion of the study, or who did not agree that the subject and his or her spouse should take strict contraceptive measures (condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, etc.) during the study period and within 1 year after completion of the study;
15. Volunteers judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Chinese males, aged 18-45 years old (inclusive)
Enrollment: 6 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Mass balance | From the start of administration to 240 h after administration
  Percentage of cumulative drug excretion of [14C]HSK21542 on biological pecimens(urine and faeces) accounting for total radiation drug dose.

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC0-t, AUC0-∞) | From the start of administration to 240 h after administration
  Pharmacokinetic Measures
Peak concentration (Cmax) | From the start of administration to 240 h after administration
  Pharmacokinetic Measures

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — Medical Ethics Committee of the First Affiliated Hospital of soochow University
Locations (1):
- f the First Affiliated Hospital of soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan JJ, Bian YC, Ma S, Chen W, Zhang FY, Zhang H, Miao LY. Pharmacokinetics, Mass Balance and Metabolism of [14C]HSK21542, a Novel Kappa Opioid Receptor Agonist, in Humans. Eur J Drug Metab Pharmacokinet. 2023 Nov;48(6):723-731. doi: 10.1007/s13318-023-00858-0. Epub 2023 Oct 13. PMID 37833493